CLINICAL TRIAL: NCT02954497
Title: Pumps for Kids, Infants, and Neonates
Acronym: PumpKIN
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Jarvik Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: C01367
Record Dates: First submitted 2016-10-31; First posted 2016-11-03 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2022-11

CONDITIONS: Pediatric Heart Failure
Keywords: ventricular assist device; congenital heart disease; heart failure
MeSH Terms: conditions — Heart Defects, Congenital; Heart Failure

STUDY DESIGN:
Intervention Model Description: Jarvik 2015
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Jarvik 2015 Device VAD (Experimental): New, experimental continuous flow VAD
  Interventions: Device: Surgical placement of the Jarvik 2015 VAD; Procedure: Surgical Placement of Jarvik 2015 VAD

INTERVENTIONS:
Device: Surgical placement of the Jarvik 2015 VAD — The Jarvik 2015 VAD is a miniaturized, fully implantable, continuous flow left ventricular assist device.
Procedure: Surgical Placement of Jarvik 2015 VAD — Surgical Implant of the Jarvik 2015 VAD is a miniaturized, fully implantable, continuous flow left ventricular assist device.

SUMMARY:
PumpKIN is a multicenter, prospective, single-arm feasibility study; Evaluating the investigational Jarvik 2015 VAD in pediatric patients with heart failure. This feasibility trial will enroll 10 subjects at up to 7 sites in the US.

The primary objectives of this investigational device exemption (IDE) clinical investigation are to assess the feasibility of using the Jarvik 2015 in pediatric patients with severe heart failure who require mechanical circulatory support. Feasibility will be assessed by evaluating the safety profile of the Jarvik 2015 device in eligible subjects.

ELIGIBILITY:
Children must meet all of the following criteria:

1. Males and females within weight range 8 to 30 kg
2. Body surface area (BSA) 0.4 m2 to 1.0 m2
3. Cardiac Diagnosis:

   a. Standard Cardiac Anatomy : Two-ventricle circulation, including cardiomyopathy, repaired structural heart disease (e.g. anomalous left coronary artery from the pulmonary artery [ALCAPA], aortic stenosis) or acquired heart disease (e.g., myocarditis, Kawasaki disease)
4. INTERMACS Profile 1 or 2 as evidenced by one or more of the following:

   1. Inability to wean from extra-corporeal membrane oxygenation (ECMO) or other temporary circulatory support (TCS), OR
   2. Inability to wean from mechanical ventilator support, OR
   3. Inotrope-dependent, decompensated heart failure AND meet one or more of the following criteria within 48 hours prior to implant (unless otherwise noted) which is attributed to decompensated heart failure despite optimal medical therapy:

   i. Urine output <0.5 cc/kg/hour for 12hr within 48 hours ii. Creatinine level >2 times the ULN for age iii. Alanine aminotransferase (ALT) or total bilirubin result >3 times the ULN for age (either qualifies the patient) iv. Mixed venous oxygen saturation (SvO2) <55% (or arteriovenous oxygen difference of >45%) in two repeated measurements v. Acidosis: Base excess >-5 in 2 or more measurements vi. Inability to tolerate appropriate enteral calories as prescribed by a registered dietician d. Inability to ambulate freely to participate fully in age-appropriate activities of daily living (ADLs) and/or cardiac rehabilitation/physical therapy
5. LVAD support is intended for bridge-to transplant. Subject is listed for transplant or eligible (i.e., no medical or surgical contraindications) to be listed for cardiac transplant, United Network for Organ Sharing (UNOS) status 1A, or equivalent
6. Written consent of parent(s) or legally authorized representative (LAR) where appropriate.

Children must not meet any of the following exclusion criteria within 48 hours prior to device implant:

1. Known contraindication for systemic anticoagulation
2. Currently participating in an interventional trial whose protocol prevents effective application of Jarvik 2015, potentially has an independent effect on trial endpoints, or otherwise interferes with execution of the PumpKIN protocol
3. Stable inotrope dependence (INTERMACS profile 3)
4. Single ventricle anatomy
5. Presence of a mechanical heart valve
6. Unresolved malignancy
7. CPR with duration >30 consecutive minutes within 48 hours prior to device implant or CPR with uncertain neurological status prior to device implant
8. Renal dysfunction that is severe or, in the opinion of the investigator, irreversible
9. Hepatic dysfunction that is severe or, in the opinion of the investigator, irreversible
10. Severe or irreversible pulmonary dysfunction
11. ECMO use for >10 consecutive days
12. Unrepairable severe aortic insufficiency
13. Active, systemic infection unresponsive to antimicrobial therapy
14. Known cerebrovascular event within the past 30 days or uncertain neurological status
15. Severe right ventricular (RV) dysfunction or significant arrhythmia requiring treatment with an RV assist device (RVAD) (i.e., biventricular assist device)
16. Unmanageable bleeding per judgment of the investigator
17. Ventricular dysfunction that is likely to recover (e.g. myocarditis, metabolic myopathy where LV dysfunction is present solely with intermittent acidosis/crises).
18. Left ventricular end-diastolic dimension or left ventricular end-diastolic volume z score of < +2.5 end-diastolic dimension or ventricular end-diastolic volume z score of < +3.0
19. Left ventricular ejection fraction of >35%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Feasibility | 30 days or transplant/recovery (whichever comes first)
  To assess the clinical feasibility of the investigational Jarvik 2015 VAD by evaluating survival in the absence of severe neurological impairment or death, or device failure up to the clinical endpoint defined as transplant, recovery or 30 days of support
Adverse Events | 30 days or transplant/recovery (whichever comes first)
  To evaluate the protocol defined (INTERMACS version 5.0) serious adverse events on Jarvik 2015 support up to transplant, recovery or 30 days of support
Technical, surgical, and clinical milestones assessed by feasibility milestones | up to 180 days or transplant/recovery
  To describe the technical, surgical and clinical feasibility by achieving specific technical, surgical, and clinical milestones that typically accompany a successful VAD support run
Pivotal Trial continuation assessed by exploratory primary and secondary endpoints | 12-months post-explant
  To evaluate patients with respect to exploratory primary and secondary endpoints to inform the choice of appropriate primary and secondary endpoints for the pivotal trial.

SECONDARY OUTCOMES:
Incidence of Adverse Events per patient days of VAD support | 180 days post-implant
  The incidence rate of protocol-defined AEs (INTERMACS, version 5) per patient-day of VAD support up to the first 180 days post-implant.
Incidence of Adverse Events related to device | 180 days post-implant
  Incidence rate of protocol-defined AEs possibly, probably, or definitely related to the device per day of mechanical circulatory support, up to the first 180 days post-implant.
Neurological dysfunction | 180 days post-implant
  The incidence of new neurological dysfunction up to 180 days post-implant.
Pediatric Stroke Outcome Measure Neurological Exam (PSOM-NE) score (0 - 10 scale, higher = worse outcome) | 180 days and 12 months post-explant
  Pediatric Stroke Outcome Measure-Neurological (PSOM-NE) score measured at 180 days post-implant or immediately prior to explant, and at 12 months post-explant.
King's Outcome Scale for Childhood Head Injury score (0 -5 scale, higher = worse outcome) | 180 days and 12 months post-explant
  King's Outcome Scale for Childhood Head Injury (KOSCHI) score measured at 180 days post-implant or immediately prior to explant, and at 12 months post-explant.
Pediatric Stroke Recurrence and Recovery Questionnaire score (0 -10 scale, higher = worse outcome) | 180 days and 12 months post-explant
  Pediatric Stroke Recurrence and Recovery Questionnaire (RRQ) measured at 180 days post-implant or immediately prior to explant, and at 12 months post-explant.
Vineland Adaptive Behavior Scales score (scoring and scale different by domain) | 12 months post-explant
  Vineland Adaptive Behavior Scales (VABS II) measured at 12 months post-explant.
Pediatric Quality of Life score (0-4 scale per domain, higher = worse outcome) | 12 months post-explant
  PedsQL20 measured at 180 days post-implant or immediately prior to explant and 12 months post-explant.
Ventricular Assist Device Quality of Life score (scoring and scale different per question) | 30 days, 90 days, 12 months post-explant
  VAD QL measured at 30 and 90 days post-implant, and every 90 days thereafter, while on Jarvik 2015 VAD support.
Paralytics discontinuation | 12 months post-explant
  Time to discontinuation of paralytics
TPN discontinuation | 12 months post-explant
  Time to discontinuation of total parenteral nutrition (TPN)
Extubation | 30 days post-implant
  Time to extubation
Inotropic agents | 12 months post-explant
  Time to discontinuation of inotropic agents
Sedation | 30 days post-implant
  Time to discontinuation of sedation such that subject is alert and interactive (e.g., engaging in age-appropriate play).
MRI | 12 months post-explant
  Brain Magnetic Resonance Imaging (MRI) performed 12 months post-explant to assess for clinically silent neurologic injuries.
Survival in absence of severe neurological impairment | 180 days or tranplant/recovery (whichever comes first)
  Overall survival in the absence of a severe neurologic impairment and in the absence of device failure at 180 days following VAD implant and meeting any of the following outcomes: Survival to induction of anesthesia for cardiac transplant surgery, Recovery (removal of VAD and alive at 30 days post-explant), Survival at 180 consecutive days of VAD support
Overall survival in the absence of device failure | 180 days or tranplant/recovery (whichever comes first)
  Overall survival in the absence of device failure but without regard for neurologic status, meeting any of the following outcomes: Survival to induction of anesthesia for cardiac transplant surgery, Survival to recovery (removal of Jarvik 2015 VAD and alive at 30 days post-explant), Survival at 180 consecutive days of Jarvik 2015 VAD support
Survival at 30 days post-implant | 30 days post-implant
  Survival at 30 days post-implant
Survival at 180 days post-implant | 180 days post-implant
  Survival at 180 days post-implant
Survival at 12 months post-explant | 12 months post-explant
  Survival at 12 months post-explant
Time to pump failure | device explant
  Time to first pump failure
Incidence rate of pump failure | device explant
  Incidence rate of pump failures
Time to first pump exchange | device explant
  Time to first pump exchanges
Incidence rate of pump exchange | device explant
  Incidence rate of pump exchanges
Creatinine level | 180 days or immediately prior to explant
  Proportion of subjects with a creatinine level below the ULNULN
ALT level | 180 days or immediately prior to explant
  Proportion of subjects with an alanine aminotransferase (ALT) level below the ULNULN

CONTACTS AND LOCATIONS:
Overall Officials: William T Mahle, MD, Study Chair — Children's Hospital of Atlanta, Emory University School of Medicine
Locations (7):
- United States (7):
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Medical Center - Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Limited use data set will be made available through NHLBI after the conclusion of the trial.